CLINICAL TRIAL: NCT06446297
Title: Investigating the Experiences of Generational Diversity Within the Medical Profession of the National Health Service: An Exploratory Study Amongst Post-Graduate Doctors in Training
Brief Title: Generational Diversity in the Medical Profession
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: University of Plymouth (Other); Health Education England, Wessex (Other)
Responsible Party: Sponsor
Other Study IDs: 330463
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Generation Gap; Generations; Intergenerational Relations
Keywords: Generation; Generation Gap; Generational Diversity; Intergenerational workforce
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Generational X: Date of Birth (DOB) categorisation of Generation X: 1st January 1965 - 31st December 1980.
  PGDiTs recruited from the local hospital will be stratified into generational groups according to their date of birth. The investigators anticipate on having approximately two focus groups per generation.
  Interventions: Other: Focus Group.
- Generation Y: DOB categorisation of Generation Y: 1st January 1981 - 31st December 1995. PGDiTs recruited from the local hospital will be stratified into generational groups according to their date of birth. The investigators anticipate on having approximately two focus groups per generation.
  Interventions: Other: Focus Group.
- Generation Z: DOB categorisation of Generation Z: 1st January 1996 - 31st December 2010. PGDiTs recruited from the local hospital will be stratified into generational groups according to their date of birth. The investigators anticipate on having approximately two focus groups per generation.
  Interventions: Other: Focus Group.

INTERVENTIONS:
Other: Focus Group. — Participants in each focus group will attend a face-to-face (or virtual) meeting that lasts approximately 90 minutes. This will be composed of a briefing period, interview period supported and guided by an interview schedule and finishing with a debrief period. The same process will be followed if individual semi-structured interviews are undertaken.

SUMMARY:
The purpose of this work is to investigate how post-graduate doctors in training (PGDiTs) experience generational diversity with their colleagues in the workplace. The investigators want to explore and understand how PGDiTs perceive and experience generational diversity in the workplace and look into where these differences between generations could come from.

The research team wants to do this by running focus groups. These focus groups would be made up of PGDiTs that are working within one hospital. The doctors will be split into the different generations (i.e. generation X, Y and Z). A set list of questions will be used to prompt and guide the focus group conversations. Each focus group will be audio-recorded using an electronic device and then analysed with the aid of computer software. The investigators will then generate themes from the data and use this to create an overall story of the data.

It is hoped that this research can help inform supervisors and employers of the impact of generational diversity on on PGDiTs. This may be used to help develop ways of improving working relationships for PGDiTs with their supervisors and employers.

DETAILED DESCRIPTION:
The different generations and the differences between them has provided considerable interest within the media, organisations and academia. A new generation entering the workforce often prompts new conversations about the differences between all generations. Investigating these generational differences has been attempted with mixed levels of success. Some organisations have made suggestions to overcome these generational differences and improve the workplace environment. The National Health Service (NHS) is one of the largest organisations in England, but very limited research investigating generational differences in the NHS has been done.

Post-graduate doctors in training (PGDiTs) are doctors working in recognised training schemes in the NHS. These doctors range from newly qualified doctors working in the Foundation Year training scheme to doctors with over a decade of experience working in their specialist areas. The last two decades have witnessed a number of changes to these doctors' working lives, some positive and some negative. The impact of generational diversity amongst these doctors has not been looked at. These doctors are likely to experience generational diversity with their supervisors, who may have completed training several years previously.

Research Question and Objectives:

The investigators want to answer the question: how do PGDiTs experiences generational diversity in an NHS hospital? The objectives are to explore and understand the concept, perceptions, experiences and sources of generational diversity of PGDiTs working in the NHS.

Study Design:

This study will involve the use of qualitative semi-structured face-to-face focus groups to explore and understand the concept, perceptions, experiences and sources of generational differences amongst PGDiTs. The focus groups will be stratified according to the generational cohorts of the participants. The study methodology supporting our study design is pragmatic with components of grounded theory and interpretative phenomenological analysis being used. Inductive thematic analysis will be used as our method of data analysis.

Contingency arrangements are also available for certain situations. In the event that face-to-face group meetings are not practically possible due to logistical reasons then virtual meetings will be arranged. If insufficient numbers of participants are recruited to conduct focus groups then semi-structured interviews will be conducted.

The consent process has been directed by the HRA's consent and participation guidance. Prior to participating in the study, all participants must electronically agree via email. All potential participants will receive an electronic copy of the informed consent form and participant information sheet (PIS) and be provided with an opportunity to ask any question of the research team. This opportunity for questions can occur via phone call, email or as a face-to-face meeting. Participants will be asked via email to confirm their participation in the research study and willingness to complete the consent form. On the day of the focus group, each participant will be provided with a printed version of the informed consent form and asked to complete it.

Data analysis:

Each focus group will be directed primarily by the interview schedule. Each focus group will be electronically audio-recorded and subsequently transcribed. Data analysis will be conducted using thematic analysis with the generation of codes and themes. Data analysis software will be used for thematic analysis.

ELIGIBILITY:
The following criteria must all be met to permit inclusion in the research study:

* Any medically qualified healthcare professional with a General Medical Council (GMC) registration number, AND
* Currently working in a recognised training programme in the Southwest (i.e. foundation year training, integrated medical training, core surgical training, acute care common stem training, higher specialty training), AND
* Currently based at University Hospitals Plymouth (UHP), AND
* Consents to being interviewed and recorded for the purposes of the study.

An individual will be excluded from the study if any of the following criteria are met:

* Any medically qualified professional with a GMC registration number that is not currently enrolled within a recognised training programme at UHP, OR
* any medical professional working outside of UHP, OR
* employed as an Allied Health Professional, Advanced Clinical Practitioner, Advanced Critical Care Practitioner or Physician Associate will not be eligible for inclusion in the study, OR
* any individual eligible for inclusion into the study that does NOT consent to being interviewed OR recorded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants must a postgraduate doctor-in-training working within a recognised training programme in the Southwest of England and currently based at University Hospitals Plymouth NHS Trust. This will range from newly qualified doctors that are working within the foundation programme to doctors that are working in higher specialty training programmes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Thematic Analysis | 4 months.
  Qualitative data analysis will be conducted using thematic analysis to generate a number of codes and themes from the transcripts generated from focus groups and semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Boissaud-Cooke, MBChB MRCS, Principal Investigator — NHS England South West, University Hospitals Plymouth NHS Trust

IPD SHARING:
Plan to Share IPD: No
Data will be collected and retained in accordance with the United Kingdom Data Protection Act (2018) and the General Data Protection Regulation (GDPR, 2016).
  Given the nature of the data that is collected, we do not plan on making individual participant data available to other researchers. The final data set will be anonymised and shared with the relevant members of the study research team only. The anonymised data (i.e. anonymised transcripts and the thematically analysed data) will be archived by the Research and Development Department of University Hospitals Plymouth NHS Trust (Plymouth, United Kingdom).
  The investigators will only report or publish non-identifiable and anonymised sections of individuals' transcripts.

REFERENCES:
- [Derived] Boissaud-Cooke MA, Yatham S, Hardy LJ, Higginson I, Thurlow J, Schofield P. Generational diversity among postgraduate doctors in training in the NHS: protocol for a qualitative study. BMJ Open. 2025 May 7;15(5):e097320. doi: 10.1136/bmjopen-2024-097320. PMID 40341154